CLINICAL TRIAL: NCT03454919
Title: A Phase II Clinical Study on Efficacy of Palbociclib in Advanced Acral Melanoma With Cell Cycle Gene Aberrations
Brief Title: Efficacy of Palbociclib in Advanced Acral Melanoma With Cell Cycle Gene Aberrations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Kiang Wu Hospital (Other)
Responsible Party: Principal Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003
Record Dates: First submitted 2018-02-12; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Palbociclib (Other): single arm
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Drug: palbociclib; ibrance; Pfizer Inc，New York，NY Schedule: Recommended initial dosage 125mg/d，3 weeks on, 1 week off. If grade 3 or 4 adverse events occur during treatment，dosage could be reduced to 100mg/d, even 75mg/d.
  Duration: till disease progression or drug intolerance.
  Other Names: ibrance

SUMMARY:
It is a prospective, phase II, open-labeled, clinical trial aimed to determine the efficacy of palbociclib in advanced melanoma patients who bear gene aberrations in cell cycle pathways [including CDK4 amplification and/or CCND1 amplification and/or P16 (CDKN2A) loss]. Fifteen patients, if there is a response then further 45 patients will be enrolled. Totally 60 subjects with known above-mentioned gene aberrations who comply with the inclusion and exclusion criteria will be enrolled, their serum samples (at the time of the first administration of palbociclib and every 4 weeks afterwards) will be collected. Palbociclib will be given in the dose of 125 mg orally qd d1-21 every 28 days, unless disease progression or intolerance. All patients will be evaluated for the response to palbociclib by Response Evaluation Criteria in Solid Tumors (RECIST) at baseline. The standard radiographic imaging (CT scans) will be performed every 4 weeks until the end of treatment.

DETAILED DESCRIPTION:
This study is to evaluate efficacy of palbociclib in advanced acral melanoma patients with gene aberrations in cell cycle pathways [including CDK4 amplification and/or CCND1 amplification and/or P16 (CDKN2A) loss].

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years;
2. ECOG performance status 0 or 1 before treatment;
3. Metastatic melanoma or unresectable acral melanoma;
4. Histologically confirmed melanoma.
5. Bearing gene aberrations in cell cycle pathways [including CDK4 amplification and/or CCND1 amplification and/or P16 (CDKN2A) loss].;
6. Anticipated life expectancy ≥ 3 month;
7. Adequate organ function, defined as following criteria:

   1. Platelets 75 x 109/L, Hemoglobin 9.0 g/dL, Absolute Neutrophils(ANC) ≥ 1.5x109/L;
   2. Serum bilirubin ≤ 1.5*upper limit of normal (ULN) (could be ignored in the case of Gilbert's syndrome) ，Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 1.5 * ULN;
   3. Blood urea nitrogen (BUN) ≤ 1.5 * ULN, serum creatinine (Cr) ≤ 1.5 * ULN.
   4. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (LLN) as assessed by multigated acquisition (MUGA) scan or echocardiography;
   5. QTc interval: male < 450msec, female < 470msec (via Fridericia method)
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
9. Written informed consent signed.

Exclusion Criteria:

1. Previous or current administration of any kind of CDK4/6 inhibitors;
2. Administration of any other anti-tumor therapy (including but not limited to radiotherapy, chemotherapy, endocrinal therapy, surgery, molecular targeted therapy, immunotherapy or biological therapy) 4 weeks before inclusion; administration of mitocycin or nitrosamines 8 weeks before inclusion;
3. Non-treated brain metastasis (treatment controlled stable brain metastasis judged by investigators excluded);
4. Presence of third space fluid that cannot be controlled by drainage or other means (i.e. pleural effusion or ascites);
5. Long-term steroid therapy required;
6. Uncorrectable hypokalemia or hypomagnesaemia before inclusion;
7. Concurrent administration of drugs with potential of QT interval prolongation (such as antiarrhythmic drugs);
8. Allergies or previous history of severe allergies;
9. Active HBV or HCV infection (HBV viral copy number ≥ 104 copies/ml, HCV ≥ 103 copies/ml);
10. NCICTCAE Grade 2 toxicity before inclusion;
11. Diagnosed as any second primary malignant tumor in 5 years before inclusion;
12. Following conditions occur in the 6 months before drug administration: severe/ unstable angina pectoris, myocardial infarction, congestive heart failure with symptoms, cerebrovascular accident, including transient ischemic attack, pulmonary embolism, ≥ grade II renal dysfunction, and other severe diseases that investigators judged to be unsuitable for this trial;
13. Administration of potent CYP3A4 inhibitors in 7 days before inclusion , or administration of potent CYP3A4 inhibitors in 12 days before randomization ；
14. NCICTCAE Grade ≥ 2 Active arrhythmias;
15. Hypertension, defined as systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg，and cannot be controlled by medication;
16. No recommendation to receive >2 mg Warfarin treatment in 2 weeks before study beginning. It is permitted to use low dose Warfarin(<2 mg／3day) to prevent deep venous thrombosis. Low molecular weight heparin (fractionated) or aspirin are also allowed;
17. Existence of any disease affecting drug absorption, including but not limited to: no ability to swallow oral medications, active inflammatory bowel disease, partial or complete obstruction, partial or total gastrectomy, extensive bowel resection or chronic diarrhea;
18. Known infection of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or congenital immune deficiency diseases, organ transplantation history;
19. Pregnancy, breastfeeding, childbearing age female who is reluctant to take effective contraceptive measures throughout trial period. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 7 days before randomization and at first day of every cycle on visit.
20. Other severe acute or chronic physiological or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
21. Current treatment on another clinical trial. Supportive care or non-therapeutic clinical trials are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  complete and partial response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival
6-month PFS rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  6-month PFS rate
AE | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  adverse events

REFERENCES:
- [Derived] Mao L, Dai J, Cao Y, Bai X, Sheng X, Chi Z, Cui C, Kong Y, Zhang Y, Wu L, Wang X, Tang B, Lian B, Yan X, Li S, Zhou L, Wei X, Li C, Qi Z, Si L, Guo J. Palbociclib in advanced acral melanoma with genetic aberrations in the cyclin-dependent kinase 4 pathway. Eur J Cancer. 2021 May;148:297-306. doi: 10.1016/j.ejca.2021.02.021. Epub 2021 Mar 23. PMID 33770575